CLINICAL TRIAL: NCT00002634
Title: N7: EVALUATION OF MAXIMAL CHEMOTHERAPY DOSE INTENSITY PLUS MONOCLONAL ANTIBODY 3F8 IN THE TREATMENT OF NEUROBLASTOMA
Brief Title: Chemotherapy, Radiation Therapy, Immunotherapy, and Bone Marrow Transplantation in Treating Patients With Neuroblastoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Purpose: Treatment
Other Study IDs: 94-011; CDR0000064084 (Registry Identifier: PDQ (Physician Data Query)); MSKCC-FDR001041; NCI-V95-0622
Record Dates: First submitted 1999-11-01; First posted 2004-08-23 (Estimated); Last update posted 2013-07-03 (Estimated); Status verified 2013-07

CONDITIONS: Neuroblastoma
Keywords: localized resectable neuroblastoma; regional neuroblastoma; disseminated neuroblastoma; recurrent neuroblastoma; localized unresectable neuroblastoma
MeSH Terms: conditions — Neuroblastoma | interventions — Filgrastim; humanized 3F8 anti-GD2 monoclonal antibody; Cisplatin; Cyclophosphamide; Doxorubicin; Etoposide; Mesna; perfosfamide; Vincristine

INTERVENTIONS:
Biological: filgrastim
Biological: monoclonal antibody 3F8
Drug: cisplatin
Drug: cyclophosphamide
Drug: doxorubicin hydrochloride
Drug: etoposide
Drug: mesna
Drug: perfosfamide
Drug: vincristine sulfate
Procedure: autologous bone marrow transplantation
Procedure: in vitro-treated bone marrow transplantation
Radiation: low-LET cobalt-60 gamma ray therapy
Radiation: low-LET photon therapy
Radiation: radioisotope therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining chemotherapy with bone marrow transplantation may allow the doctor to give higher doses of chemotherapy drugs and kill more tumor cells. Radiation therapy uses high-energy x-rays to damage tumor cells. Monoclonal antibodies can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells.

PURPOSE: Phase II trial to study the effectiveness of combining chemotherapy, radiation therapy, immunotherapy, and bone marrow transplantation in treating patients with neuroblastoma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Improve the complete remission rate and progression-free survival and reduce the relapse rate of patients with poor-risk neuroblastoma using intensive multimodality therapy: cyclophosphamide/doxorubicin/vincristine and cisplatin/etoposide, external-beam radiotherapy, and surgery (when feasible), followed by radioimmunotherapy with iodine I 131 labeled monoclonal antibody 3F8 followed by autologous bone marrow transplant and immunotherapy with unlabeled 3F8. II. Identify biologic and clinical prognostic factors that may guide future modifications in treatment approaches for this malignancy.

OUTLINE: Patients are stratified by prior therapy (yes vs no). Patients undergo surgery either at diagnosis or after at least 4 courses of chemotherapy, then possibly again after completion of chemotherapy. Patients receive cyclophosphamide IV over 6 hours on days 1-2, and doxorubicin IV and vincristine IV over 72 hours on days 1-3 for courses 1, 2, 4, and 6. Cisplatin IV over 1 hour on days 1-4 and vincristine IV over 2 hours on days 1-3 are administered as courses 3, 5, and 7. Courses are administered every 16-21 days. Autologous bone marrow is collected after 3 courses of chemotherapy providing marrow is negative for tumor cells. Patients undergo radiotherapy after the completion of chemotherapy. Radiotherapy is administered twice a day for 7 days. Patients then receive iodine I 131 labeled monoclonal antibody 3F8 (MOAB 3F8) on day -5 and again on days 1-5. Autologous bone marrow is reinfused on day 5 and filgrastim (G-CSF) is administered IV or subcutaneously beginning day 6. Patients who do not develop HAMA or an allergy to mouse proteins receive unlabeled MOAB 3F8 IV over 1.5 hours, 5 days a week for 2 weeks. Treatment repeats every 1-2 months for up to 4 courses. Patients are followed every month for 2 years, every 3 months for 1 year, then annually thereafter.

PROJECTED ACCRUAL: Up to 45 newly diagnosed patients will be accrued for this study within 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Neuroblastoma diagnosed in accordance with the International Neuroblastoma Staging system: Histologic confirmation at MSKCC OR Elevated urinary catecholamines plus tumor cells/clumps in bone marrow Stage IV or Stage II/III with more than 10 copies of N-myc proto-oncogene per tumor cell

PATIENT CHARACTERISTICS: See General Eligibility Criteria

PRIOR CONCURRENT THERAPY: Prior therapy allowed -Patient Characteristics-- Age: Over 1 year at diagnosis Performance status: Not specified Hematopoietic: Absolute neutrophil count at least 500/mm3 (except for cases of bone marrow infiltration by tumor) Platelet count at least 100,000/mm3 (except for cases of bone marrow infiltration by tumor) Hepatic: Not specified Renal: Not specified Other: No history of allergy to mouse proteins Human antimouse antibodies (HAMA) less than 1,000 U/ml (with prior exposure to murine antibodies)

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 1995-02; Primary Completion 2004-09 (Actual); Study Completion 2004-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nai-Kong V. Cheung, MD, PhD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Background] Cheung NV, Kushner BH, LaQuaglia MP, et al.: Anti-Gd2 monoclonal antibody (MOAB) 3F8-targeted therapy and dose intensity for children (1 yr of age) with stage 4 neuroblastoma (NB): key variables in sequential protocols at Memorial Sloan Kettering Cancer Center (MSKCC). [Abstract] Proceedings of the American Society of Clinical Oncology 19: A-2305, 2000.